CLINICAL TRIAL: NCT03635476
Title: Survey of Lifelong Food and Nutrition Assistance (LIFANA) in Stroke Patients and Caregivers - Cereneo Schweiz AG (Center for Neurology and Rehabilitation)
Brief Title: Survey of Lifelong Food and Nutrition Assistance (LIFANA) in Stroke Patients and Caregivers
Status: Completed | Type: Observational
Sponsor: Cereneo AG (Industry)
Collaborators: cereneo Institute for Interdsciplinary Research (cefir) (Unknown)
Responsible Party: Principal Investigator, Krizia Ferrini, Nutritional Specialist, Cereneo AG
Other Study IDs: LIFOCUS
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Relatives; Diet Modification
Keywords: Stroke Rehabilitation; Personalized Nutrition; Mobile-Health; Stroke
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative interview study — The group in question is part of a research program aimed at developing and evaluating the LIFANA Nutrition Solution, a meal planning recommended system, which suggests meals based on the user's personal profile. This may include general preferences, such as culture, taste, and budget, but more importantly automated and personalised nutritional recommendations based on advice provided by professional nutritionists and allergists.
  Other Names: Survey

SUMMARY:
Many elderly suffer from nutritional problems that can cause (or can be caused by) a number of complications such as weakened immune systems and chronic health conditions (diabetes type 2, high blood pressure, cardiovascular diseases or even osteoporosis).

Through appropriate adjustments in the diets, on the basis of nutritional advice, the burden of established diseases as well as the risks of developing further conditions can be diminished. The goal of our proposed project LIFANA is to develop and evaluate the LIFANA Nutrition Solution to support healthy nutrition.. This may include general preferences, such as culture, taste, and budget, but more importantly automated and personalised nutritional recommendations based on advice provided by professional nutritionists and allergists. This is a national project co-funded by the European Union.

One of the activities of the project is to collect information through a survey with patients. These questions will contribute to creating solutions that can explore the perspectives of patients.

DETAILED DESCRIPTION:
Patients will be approached in the clinic by a neurologist and health care professionals. The questionnaire will take place at cereneo. The group will consist of 25 participants and last between 1h. The Survey will be conducted by a clinician who will take notes. Semi-structured discussion guide will be used. With regard to the communication, the moderator will identify factors that will influence communication in a positive or negative way.

The health professionals will perform content analyses on the transcripts; the schema of categories will be oriented towards the research questions, using open questions, directly addressing quiet participants, and handling the discussion guide in a flexible way.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients undergoing rehabilitation
* caregivers of stroke patients

Exclusion Criteria:

* Severe aphasia
* Severe cognitive deficits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: stroke patients undergoing rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
User Needs | 1 day/session
  The primary endpoint of this study is to explore the perspectives of patients through appropriate adjustments of focus group questions on user needs for managing nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Krizia Ferrini, PhD, Principal Investigator — cereneo Schweiz AG | center for neurology & rehabilitation; Doris Mösinger, MSc, Study Chair — cereneo Schweiz AG | center for neurology & rehabilitation; Leopold Zizlsperger, MD, Study Director — cereneo Schweiz AG | center for neurology & rehabilitation
Locations (1):
- cereneo Schweiz AG, Vitznau, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No